CLINICAL TRIAL: NCT02997098
Title: Longitudinal Outcomes in Hepatic Resection
Status: Withdrawn | Type: Observational
Why Stopped: Study design changed to clinical database only with no research question to be studied.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00078618
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Liver Diseases; Surgery
Keywords: Hepatectomy
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing hepatectomy: Patients undergoing hepatectomy, or liver resection, for a non-transplant indication.

SUMMARY:
This observational registry of patients undergoing liver surgery collects patients both retrospectively and prospectively. Patients undergoing liver resection for any non-transplant indication will be evaluated for clinical outcomes (such as surgical complications, survival, and disease progression) based on clinical and patient factors (like indication, age, and other treatments for the disease).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring liver resection

Exclusion Criteria:

* Patients under the age of 18 years
* Patients undergoing liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver resection for non-transplant indications.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2037-05 (Estimated); Study Completion 2037-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years

SECONDARY OUTCOMES:
Disease-free survival | 10 years
Surgical-site infection | 3 months
Postoperative bleeding | 3 months
Blood clot | 3 months
Use of other therapy | 5 years
  e.g., antibiotics in liver abscess, chemotherapy in liver cancer
Operative time | 1 day
Intraoperative blood loss | 1 day
Number of segments resected | 1 day
  If applicable

CONTACTS AND LOCATIONS:
Overall Officials: Sabino Zani, MD, Principal Investigator — DUHS
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No